CLINICAL TRIAL: NCT01650233
Title: Improving Wellness for Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NA_00028889
Record Dates: First submitted 2012-07-20; First posted 2012-07-26 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Stress-exposed Urban Male Youth
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness-based stress reduction (Experimental): The mindfulness-based stress reduction (MBSR) program was previously adapted for urban youth and here further adapted to 12 weekly 50-minute classes for use in school.
  Interventions: Behavioral: Mindfulness-based stress reduction
- Healthy Topics (Placebo Comparator): An age-appropriate health education curriculum was used as a non-specific group comparison for the MBSR program to control for the effects of: positive adult instruction, interactive peer group instruction, learning new material, group size and location, time, and attention.
  Interventions: Behavioral: Mindfulness-based stress reduction

INTERVENTIONS:
Behavioral: Mindfulness-based stress reduction

SUMMARY:
This study assesses the impact of a mindfulness-based stress reduction program compared with a health education program for urban middle-school male youth on outcomes of psychological symptoms, coping, stress, sleep, and behavior.

ELIGIBILITY:
Inclusion Criteria:

* 7th or 8th graders at St. Ignatius Loyola Academy in 2009-2010 academic year.
* Parent/guardian consents
* Student assents

Exclusion Criteria (as assessed by school staff):

* significant psychopathology
* significant developmental delay
* significant substance abuse with behavioral consequences
* significant behavioral problems
* foster care due to consent restrictions)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-08; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
psychological symptoms | 6 months
  Psychological symptoms assessed include anxiety, hostility, and depression.
coping | 6 months
  Coping assessed includes rumination and typically positive and negative coping approaches.

SECONDARY OUTCOMES:
Sleep | 6 months
  Sleep was measured using diary and actigraphy.
stress | 6 months
  Stress was measured using self-report and salivary cortisol.

OTHER OUTCOMES:
Behavior | 6 months
  Assessed by teacher-rated behavior ratings.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Ignatius Loyola Academy, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Sibinga EM, Perry-Parrish C, Chung SE, Johnson SB, Smith M, Ellen JM. School-based mindfulness instruction for urban male youth: a small randomized controlled trial. Prev Med. 2013 Dec;57(6):799-801. doi: 10.1016/j.ypmed.2013.08.027. Epub 2013 Sep 9. PMID 24029559